CLINICAL TRIAL: NCT01703312
Title: A Randomized, Double-blind, Placebo- and Comparator-controlled Study Evaluating the Effect of Multiple Doses of QGE031 Compared to Omalizumab in Asthma Induced by Allergen Bronchial Provocation
Brief Title: A Study Evaluating the Efficacy of QGE031 Compared to Omalizumab in Patients With Allergic Asthma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQGE031B2203
Record Dates: First submitted 2012-10-05; First posted 2012-10-10 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Allergic Asthma
Keywords: Allergies, asthma, IgE
MeSH Terms: conditions — Hypersensitivity; Asthma; Epilepsy, Idiopathic Generalized | interventions — ligelizumab; Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- QGE031 (Experimental): During the 10-week treatment period, participants will receive a dose of study drug subcutaneously once every two weeks (total of six doses). Three dose levels of QGE031 will be offered during the study: low, medium, and high. Participants will be randomized to receive one of these dose levels for all dosing visits.
  Interventions: Drug: QGE031
- omalizumab (Active Comparator): During the 10-week treatment period, participants will receive a dose of study drug subcutaneously once every two weeks (total of six doses) or once every four weeks (total of three doses). The dose that a participant receives will depend upon the participant's body weight and IgE level; dosage will be determined based upon local omalizumab dosing charts.
  Interventions: Drug: omalizumab
- placebo (Placebo Comparator): During the 10-week treatment period, participants will receive a dose of study drug subcutaneously once every two weeks (total of six doses).
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: QGE031 — Drug administered by subcutaneous injection
  Arms: QGE031
Drug: omalizumab — Drug administered by subcutaneous injection
  Arms: omalizumab
Drug: placebo — Drug administered by subcutaneous injection
  Arms: placebo

SUMMARY:
This study will evaluate the efficacy of QGE031 compared to omalizumab in patients with allergic asthma. Each treatment's effect in changing the concentration of inhaled allergen that is required to elicit a 15% fall in the forced expiratory volume in one second (FEV1) at 12 weeks compared to baseline will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Adult patients 18 to 65 years

Positive skin prick test to one or more common airborne allergens

Presence of airway hyperresponsiveness documented by a provocative concentration of methacholine causing a 20% fall in FEV1 (PC20 FEV1) of less than or equal to 16 mg/mL

Presence of an early asthmatic response demonstrated by an allergen challenge at screening and including a 15% fall in the FEV1

Patients with a body weight and total IgE in a range specified by local country prescribing information for omalizumab

Exclusion Criteria:

Pregnant or nursing (lactating) women

Women of child-bearing potential unless they are using a highly effective method of birth control (as further defined in the study protocol)

Smokers

Patients with poorly controlled asthma or patients who have had an asthma exacerbation within the past year

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in the concentration of inhaled allergen that elicits a 15% fall in the forced expiratory volume in one second (FEV1) | Baseline, 12 weeks

SECONDARY OUTCOMES:
Change in the concentration of inhaled allergen that elicits a 15% fall in the forced expiratory volume in one second (FEV1) following treatment with placebo and various doses of QGE031 | Baseline, 12 weeks
QGE031 blood concentrations | 24 weeks
Number of participants with adverse events or other safety concerns | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Canada (6):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Ste-Foy, Quebec
  - Novartis Investigative Site, Saskatoon, Saskatchewan
  - Novartis Investigative Site, Vancouver
- Novartis Investigative Site, Stockholm, Sweden